CLINICAL TRIAL: NCT00294398
Title: Inhaled Corticosteroids After a Pediatric Emergency Visit for Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2005-8-4458
Record Dates: First submitted 2006-02-20; First posted 2006-02-22 (Estimated); Results first posted 2015-04-24 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-04

CONDITIONS: Asthma
Keywords: Asthma, Controller Medications
MeSH Terms: conditions — Asthma | interventions — Budesonide; Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Asthma ED Discharge Therapy (Other): Standard asthma therapy including oral corticosteroids, albuterol, education and discharge instructions.
  Interventions: Other: Standard Asthma ED Discharge Therapy
- ICS Prescription + Standard Asthma ED Discharge Therapy (Experimental): Subjects are given a prescription for a 30 day supply of an inhaled corticosteroid based on age:
  1-4 year olds Budesonide 0.5mg via nebulizer once daily; 5-11 year olds Fluticasone propionate 44mcg 2 puffs via spacer twice daily; 12-18 year olds Fluticasone propionate 110mcg 2 puffs via spacer twice daily
  Interventions: Other: ICS Prescription + Standard Asthma ED Discharge Therapy

INTERVENTIONS:
Other: ICS Prescription + Standard Asthma ED Discharge Therapy — Subjects are given a prescription for a 30 day supply of an inhaled corticosteroid based on age:
  1-4 year olds Budesonide 0.5mg via nebulizer once daily; 5-11 year olds Fluticasone propionate 44mcg 2 puffs via spacer twice daily; 12-18 year olds Fluticasone propionate 110mcg 2 puffs via spacer twice daily
  Other Names: Budesonide; Fluticasone propionate; Pulmicort; Flovent
  Arms: ICS Prescription + Standard Asthma ED Discharge Therapy
Other: Standard Asthma ED Discharge Therapy — Subjects are instructed to use albuterol as needed (up to every 4 hours), may be prescribed prednisone and to follow-up with their primary doctor in 3-5 days. All view an educational video about asthma control and are provided a home nebulizer if needed.
  Other Names: Control
  Arms: Standard Asthma ED Discharge Therapy

SUMMARY:
Specific Aim:

To determine whether a prescription for Inhaled Corticosteroids (ICS) added to standard Emergency Department (ED) discharge therapy for young children with persistent asthma symptoms increases ICS use and improves symptoms and quality of life over the months following the ED visit.

Hypotheses:

In a cohort of pediatric patients with persistent asthma discharged from the ED after an acute asthma exacerbation, a prescription for ICS will:

1. Improve usage of ICS as measured by refill of a prescription within the first 2 months after the ED visit
2. Improve symptom severity at two weeks after an ED visit as measured by days of cough, wheeze, missed school, daycare or work
3. Improve patient and caregiver asthma-related quality of life during the 2 months following an ED visit measured by asthma Health Related Quality of Life (HRQL)
4. Improve asthma control at 2 months as measured by a validated asthma instrument

DETAILED DESCRIPTION:
Abstract.

Background: Asthma prevalence, emergency visits, and hospitalizations have increased substantially, especially among young children and urban populations. Although inhaled corticosteroids (ICS) are the mainstay of treatment for persistent asthma, studies have demonstrated a low rate of ICS usage and primary care provider follow-up within a month of an Emergency Department (ED) visit. Furthermore, ICS usage and adherence with National Asthma Education and Prevention Program (NAEPP) recommendations is low even for children that follow-up with their primary care physician (PCP). In addition, other studies have demonstrated frequent symptoms, activity restriction, and missed school or work during the weeks following an ED visit. Prescribing ICS at ED discharge occurs uncommonly in the United States based on surveys and reviews of current practice. Adult studies have been inconclusive and the role of ICS after a pediatric emergency visit for asthma has not been studied. This study will assess the short-term outcomes of prescribing ICS to young children with persistent asthma symptoms after an emergency visit for asthma.

Objective: To determine whether a prescription for ICS added to standard asthma ED discharge therapy to young children with persistent asthma increases adherence to NAEPP guidelines for ICS usage at 2 months follow up and improves short-term symptoms and quality of life for patient and caregiver.

Methods: Randomized control trial of children 1- 8yo of age with persistent asthma being discharged after an emergency visit for asthma. Subjects will be randomized to receive standard therapy of oral corticosteroid, albuterol, and education versus standard care plus a prescription for budesonide once daily. A questionnaire will be administered at baseline, with follow-up telephone interviews conducted at 2 weeks and 2 months. Pharmacy verification of refill of a second prescription of ICS will be the primary outcome. Asthma symptoms and quality of life will be assessed as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 12 months through 18 years
2. History of asthma defined as 2 or more prior physician visits at which bronchodilators were prescribed
3. Persistent symptoms identified by an asthma control tool based on the NAEPP Guidelines and developed and validated by a multidisciplinary team of clinicians from CHOP Allergy, Pulmonary Medicine, General Pediatrics and Emergency Medicine.
4. Treated in ED for acute asthma with plan to discharge from the ED on oral prednisone
5. Have a Primary Care Physician (PCP)

Exclusion Criteria:

1. Current hospitalization or admission to the extended day emergency care unit
2. History of pediatric intensive care admission for asthma
3. Current prescription for a controller medication such as inhaled corticosteroids (ICS), leukotriene receptor antagonists, or cromolyn
4. Contraindications to the use of routine asthma medications including beta-agonists or systemic steroids
5. Co-morbid disease: Chronic lung disease, for example cystic fibrosis; Congenital heart disease requiring surgery and/or medications; Sickle cell disease; Immunodeficiency syndromes
6. Previous enrollment in the study

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 152 (Actual)
Dates: Start 2006-03; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther M Sampayo, MD, Principal Investigator — CHOP
Locations (1):
- CHOP, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Bukstein DA, McGrath MM, Buchner DA, Landgraf J, Goss TF. Evaluation of a short form for measuring health-related quality of life among pediatric asthma patients. J Allergy Clin Immunol. 2000 Feb;105(2 Pt 1):245-51. doi: 10.1016/s0091-6749(00)90072-1. PMID 10669843
- [Background] Zorc JJ, Pawlowski NA, Allen JL, Bryant-Stephens T, Winston M, Angsuco C, Shea JA. Development and validation of an instrument to measure asthma symptom control in children. J Asthma. 2006 Dec;43(10):753-8. doi: 10.1080/02770900601031615. PMID 17169827

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened for enrollment at the Children's Hospital of Philadelphia Emergency Department (ED) between 2006 to 2009. Of the 75,000 annual ED visits in the Children's Hospital of Philadelphia ED per year, more than 6,000 of these visit represent patients with acute asthma.
Pre-assignment Details: 152 participants were enrolled and randomized between 2006 and 2009 in the Children's Hospital of Philadelphia Emergency Department.
Groups:
- Standard Asthma ED Discharge Therapy: Subjects were instructed to use albuterol as needed (up to every 4 hours), may have been prescribed prednisone and asked to follow-up with their primary doctor in 3-5 days. All viewed an educational video about asthma control and were provided a home nebulizer if needed.
- ICS Prescription + Standard Asthma ED Discharge Therapy: Subjects were given a prescription for a 30 day supply of an inhaled corticosteroid based on age:
  1-4 year olds Budesonide 0.5mg via nebulizer once daily; 5-11 year olds Fluticasone propionate 44mcg 2 puffs via spacer twice daily; 12-18 year olds Fluticasone propionate 110mcg 2 puffs via spacer twice daily
Period: Overall Study
Arm/Group | Standard Asthma ED Discharge Therapy | ICS Prescription + Standard Asthma ED Discharge Therapy
Started | 78 | 74
Completed | 57 | 48
Not Completed | 21 | 26
Not completed — Lost to Follow-up | 21 | 26

BASELINE CHARACTERISTICS:
Groups:
- Standard Asthma ED Discharge Therapy: Subjects were instructed to use albuterol as needed (up to every 4 hours), may have been prescribed prednisone and asked to follow-up with their primary doctor in 3-5 days. All viewed an educational video about asthma control and are provided a home nebulizer if needed.
- ICS Prescription + Standard ED Discharge Therapy: Subjects were given a prescription for a 30 day supply of an inhaled corticosteroid based on age:
  1-4 year olds Budesonide 0.5mg via nebulizer once daily; 5-11 year olds Fluticasone propionate 44mcg 2 puffs via spacer twice daily; 12-18 year olds Fluticasone propionate 110mcg 2 puffs via spacer twice daily
- Total: Total of all reporting groups
Arm/Group | Standard Asthma ED Discharge Therapy | ICS Prescription + Standard ED Discharge Therapy | Total
Number analyzed (Participants) | 78 | 74 | 152
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 78 | 74 | 152
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.5 (3.1) | 5.5 (4.8) | 5.0 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 36 | 66
  Male | 48 | 38 | 86
Region of Enrollment [Number; unit: participants]
  United States | 78 | 74 | 152

OUTCOME MEASURES:

1. Primary Outcome: Number of Inhaled Corticosteroid (ICS) Prescriptions Refilled (Confirmed by Primary Care Physician)
Description: Verification of a filled prescription for an ICS was completed 2 months after emergency department (ED) visit via telephone call to the pharmacy. Individual informed consent forms were faxed to the pharmacy to obtain verification that a prescription was filled. The number of subjects who filled a prescription for an ICS after the ED visit was compared between the two groups.
Time Frame: 2 months
Population: Analysis population was based on the intention to treat number at enrollment.
Measure: Number; unit: Participants
Groups:
- ICS Prescription + Standard Asthma ED Discharge Therapy:: Subjects are given a prescription for a 30 day supply of an inhaled corticosteroid based on age:
  1-4 year olds Budesonide 0.5mg via nebulizer once daily; 5-11 year olds Fluticasone propionate 44mcg 2 puffs via spacer twice daily; 12-18 year olds Fluticasone propionate 110mcg 2 puffs via spacer twice daily
Arm/Group | Standard Asthma ED Discharge Therapy | ICS Prescription + Standard Asthma ED Discharge Therapy:
Number analyzed (Participants) | 78 | 74
Participants | 18 | 32
Statistical Analysis 1: Comparison: Standard Asthma ED Discharge Therapy vs ICS Prescription + Standard Asthma ED Discharge Therapy:; Test type: Superiority or Other; p = 0.87, t-test, 2 sided

2. Secondary Outcome: Asthma-related Quality of Life
Description: Bukstein health-related quality of life instrument is an an 8-item questionnaire for measuring health-related quality of life in pediatric asthma. The daytime and nighttime symptom scales for each contain 2 items and the functional limitations scale 4 items. Prior validation studies confirm each scale's ability to detect changes at both low and high levels of functioning. The scale is scored from 0 to 100, with higher scores indicating better quality of life and lower scores translate to poorer health-related quality of life.
Time Frame: 2 months
Population: Analysis population was based on the intention to treat number at enrollment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard Asthma ED Discharge Therapy | ICS Prescription + Standard Asthma ED Discharge Therapy:
Number analyzed (Participants) | 36 | 30
units on a scale | 65 (21) | 66 (27)

ADVERSE EVENTS:
Time Frame: 2 months
Description: All subjects received follow-up telephone calls 2 weeks and 2 months following the emergency department (ED) visit.
Arm/Group | Standard Asthma ED Discharge Therapy | ICS Prescription + Standard Asthma ED Discharge Therapy
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/74
Other Adverse Events (participants affected / at risk) | 0/78 | 0/74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes